CLINICAL TRIAL: NCT03507608
Title: Randomized Trial Assessing Induction of Double Strand Breaks With Androgen Receptor Partial Agonist in Patients on Androgen Suppression
Brief Title: Assessing Induction of Double Strand Breaks With Androgen Receptor Partial Agonist in Patients on Androgen Suppression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Patrick C. Walsh Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1851; IRB00167697 (Other: JHM IRB)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide

STUDY DESIGN:
Intervention Model Description: The initial phase is a 6-patient single-arm run-in phase to test feasibility and rule out futility of the intervention. All patients within the run-in phase will receive 50mg flutamide prior to brachytherapy and prostatic biopsy. If futility is ruled out (>1 patients with DSBs on biopsy), then accrual will continue in the randomized in a 2:1 ratio (12:6 patients), for an all-trial total of 18 patients receiving flutamide vs 6 patients receiving placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- flutamide (Experimental): 50mg flutamide prior to brachytherapy and prostatic biopsy
  Interventions: Drug: Flutamide
- placebo (Placebo Comparator): placebo prior to brachytherapy and prostatic biopsy
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Flutamide — 50mg flutamide prior to brachytherapy and prostatic biopsy
  Arms: flutamide
Other: Placebo — placebo prior to brachytherapy and prostatic biopsy
  Arms: placebo

SUMMARY:
This is a prospective, single-center, two-phase study to assess the efficacy of single pulsed-dose flutamide in creating double strand breaks (DSBs) in prostate cancer within patients receiving central androgen suppression and brachytherapy.

DETAILED DESCRIPTION:
This is a prospective, single-center, two-phase study to assess the efficacy of single pulsed-dose flutamide in creating DSBs (double strand breaks) in prostate cancer within patients receiving central androgen suppression and brachytherapy. The initial phase is a 6-patient single-arm run-in phase to test feasibility and rule out futility of the intervention. All patients within the run-in phase will receive 50mg flutamide prior to brachytherapy and prostatic biopsy. If futility is ruled out (>1 patients with DSBs on biopsy), then accrual will continue in the randomized, double-blind phase. Subjects will be randomized in a 2:1 ratio (12:6 patients), for an all-trial total of 18 patients receiving flutamide vs 6 patients receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* At least one biopsy core with Gleason 7 or higher disease
* The patient has decided to undergo brachytherapy plus androgen suppression as treatment modality for his prostate cancer (with or without supplemental external beam radiation)
* Suitable volume of disease for biopsy:
* clinically palpable disease corresponding to (ipsilateral to) any involved core on biopsy
* Signed study-specific consent form prior to registration

Exclusion Criteria:

* Known hypersensitivity or allergic response to flutamide
* Severe hepatic impairment
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow up.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males with prostate cancer
Enrollment: 25 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Song, M.D., Principal Investigator — SKCCC at Johns Hopkins
Locations (1):
- SKCCC at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee E, Coulter J, Mishra A, Caramella-Pereira F, Demarzo A, Rudek M, Hu C, Han M, DeWeese TL, Yegnasubramanian S, Song DY. Induction of double-strand breaks with the non-steroidal androgen receptor ligand flutamide in patients on androgen suppression: a study protocol for a randomized, double-blind prospective trial. Trials. 2023 Dec 16;24(1):809. doi: 10.1186/s13063-023-07838-4. PMID 38104131

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants in the run-in phase received flutamide. In the second phase, additional participants were randomized, double-blind phase to receive "Flutamide" or "Placebo
Groups:
- Flutamide Run In: Single-arm run-in phase: patients within the run-in phase will receive 50mg flutamide prior to brachytherapy and prostatic biopsy. If futility is ruled out (>1 patients with DSBs on biopsy), then accrual will continue in the randomized, double-blind phase 2.
- Phase 2: DB Flutamide: Flutamide: 50mg flutamide prior to brachytherapy and prostatic biopsy
- Phase 2: DB Placebo: Placebo: placebo prior to brachytherapy and prostatic biopsy
Period: Period 1: Single-arm run-in Phase
Arm/Group | Flutamide Run In | Phase 2: DB Flutamide | Phase 2: DB Placebo
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2: Randomized, Double-blind Phase
Arm/Group | Flutamide Run In | Phase 2: DB Flutamide | Phase 2: DB Placebo
Started | 0 | 14 | 5
Completed | 0 | 14 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Run-In: 6-patient single-arm run-in phase to test feasibility and rule out futility of the intervention.
  Patients within the run-in phase will receive 250mg prior to brachytherapy and prostatic biopsy
- Flutamide: 250mg flutamide prior to brachytherapy and prostatic biopsy
  Flutamide: 250mg flutamide prior to brachytherapy and prostatic biopsy
- Total: Total of all reporting groups
Arm/Group | Run-In | Flutamide | Placebo | Total
Number analyzed (Participants) | 6 | 14 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 4 | 12
  >=65 years | 4 | 8 | 1 | 13
Age, Continuous [Mean (Full Range); unit: years] | 66 [51 to 80] | 65.86 [57 to 75] | 60.20 [53 to 75] | 64.76 [51 to 80]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male Participants | 6 | 14 | 5 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 14 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Fold-change Post Flutamide Exposure
Description: To confirm DNA double-strand breaks occur in prostate cancer tissue following pulse-dose flutamide administration in patients who are androgen suppressed. A value less than 1 indicates a decrease and a value greater than 1 indicates an increase.
Time Frame: Post Flutamide exposure up to 12 hours
Population: Patients with tumor tissue at biopsy. Patients that received Flutamide in Phase 2.
Measure: Mean (95% Confidence Interval); unit: Fold-change
Arm/Group | Flutamide | Placebo
Number analyzed (Participants) | 12 | 0
Fold-change | 5.860 [0.8680 to 8.852] |

ADVERSE EVENTS:
Time Frame: From enrollment up to 6 months
Arm/Group | Flutamide Run In | Flutamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/14 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/14 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/14 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flutamide Run In (N=6) | Flutamide (N=14) | Placebo (N=5)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — 1 patient went to emergency room post-treatment. Foley was replaced to address urinary retention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT03507608/Prot_SAP_000.pdf